CLINICAL TRIAL: NCT04943328
Title: Post Market Clinical Follow-Up (PMCF) Study to Evaluate the Performance and Safety of the Cemented TrendHip® Stem in a Prospective Follow-up Study
Brief Title: Cemented TrendHip® - Multicenter PMCF Study on Total Indications
Acronym: TRESTI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAG-O-H-2105
Record Dates: First submitted 2021-06-23; First posted 2021-06-29 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Coxarthrosis; Primary; Coxarthrosis; Post-Traumatic; Necrosis, Femur Head; Rheumatoid Arthritis; Fractures, Hip; Hip Dysplasia
Keywords: Total Hip Arthroplasty; Hip Prosthesis; Elderly Patients; Bone Cement
MeSH Terms: conditions — Osteoarthritis, Hip; Femur Head Necrosis; Arthritis, Rheumatoid; Hip Fractures; Hip Dislocation | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TrendHip® (Other)
  Interventions: Device: Total Hip Arthroplasty

INTERVENTIONS:
Device: Total Hip Arthroplasty — cemented hip arthroplasty
  Other Names: TrendHip®

SUMMARY:
This Post Market Clinical Follow-Up (PMCF) study to evaluate the performance and safety of the cemented TrendHip® stem in a prospective follow-up study with patients who underwent a hip arthroplasty with the investigational product (representative of usual clinical practice), at two follow-up examinations

ELIGIBILITY:
Inclusion: Inclusion criteria

* Patient older than 18 years.
* Patient who undergo / underwent a hip arthroplasty with cemented TrendHip® femoral stem according to the indications for implantation specified in the Instructions for Use.
* Patient not opposing participation in the study.

Exclusion: Exclusion criteria

* Patient with shortened life expectancy.
* The patient is unable to commit to the planned follow-up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2028-05-08 (Estimated)

PRIMARY OUTCOMES:
Change of functional outcome over five year follow-up period (modified Harris Hip Score) | preoperative (as available) and at two examinations during Follow-Up (1 year postop, 5 years postop)
  The modified Harris Hip Score (mHHS) as patient-reported outcome measure and evaluated one-year and five-years postoperatively. The mHHS is a validated and disease-specific instrument commonly used to assess outcomes in total hip arthroplasty. The domains covered are pain, function (gait), and functional activities.

SECONDARY OUTCOMES:
Pain Assessment | at two examinations during Follow-Up (1 year postop, 5 years postop)
  Pain will be measured with a Visual Analogue Scale (VAS), at rest and when walking on flat ground. The Visual Analog Scale (VAS) is a 10 cm line with anchor statements on the left (no pain) and on the right (extreme pain). The patients are asked to mark their current pain level on the line.
Patient satisfaction with surgery result | at two examinations during Follow-Up (1 year postop, 5 years postop)
  Patient is asked for satisfaction with surgery result with a 4-point scale: very satisfied, satisfied, unsatisfied, very unsatisfied
Survival rate (Kaplan-Meier) | at two examinations during Follow-Up (1 year postop, 5 years postop)
  The survival of the TrendHip® Total Hip Prothesis will be analyzed using the "Kaplan-Meier".
Radiological Outcome: Migration of the stem in mm | at two examinations during Follow-Up (1 year postop, 5 years postop)
  Migration of the stem is assessed in [mm] relative to postoperative x-rays
Radiological Outcome: Evaluation of bony osseointegration or conspicuous features of the stem | at two examinations during Follow-Up (1 year postop, 5 years postop)
  Bony Osseointegration or conspicuous features of the stem are assessed on anterior-posterior and lateral x-rays of the stem and will be analysed according to the zones defined by Gruen. "Charnley" and "Gruen" zones of the hip are distinct zones used in assessment of aseptic loosening in total hip joint replacements
Radiological Outcome: Heterotopic Ossification | at two examinations during Follow-Up (1 year postop, 5 years postop)
  Brooker classification divides heterotopic ossifications that form following total hip replacement to four classes. Class I: islands of bone within soft tissues around hip; Class II: bone spurs in pelvis or proximal end of femur leaving ≥1 cm between the opposing bone surfaces; Class III: bone spurs that extend from pelvis or the proximal end of femur, which reduce the space between the opposing bone surfaces to <1cm; Class IV: ankylosis of the hip on x-ray

OTHER OUTCOMES:
Rate of Adverse and Serious Adverse Events | at two examinations during Follow-Up (1 year postop, 5 years postop)
  All Adverse Events (AE) / Serious Adverse Events (SAE) observed during the follow-up examination or reported by the patient will be documented. Only those AE and SAE that could be related to the investigational product or the TrendHip® Total Hip Arthroplasty procedure are of interest.

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - St. Franziskus-Hospital, Ahlen, North Rhine-Westphalia
  - St. Vincenz Hospital Brakel, Brakel
  - St. Marien-Hospital, Mülheim
  - radprax Krankenhaus Plettenberg GmbH, Plettenberg